CLINICAL TRIAL: NCT05516212
Title: The Effect of Caffeine and Paraxantine Kinetics on Exercise Performance and Psychophysical State in Athletes After Ingestion of Mono- or Multi-ingredient Caffeine-containing Supplements
Brief Title: Caffeine Kinetics and CrossFit®-Specific Performance
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: National Science Centre, Poland (Other Government); Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Prof Dr hab., PhD, Poznan University of Physical Education
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDS2022_0003
Record Dates: First submitted 2022-06-29; First posted 2022-08-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Supplementation; Sports Nutrition; Ergogenic Support; Discipline-specific Performance
Keywords: Pre-workout supplementation; caffeine; high-intensity interval training; high-intensity functional training; performance; crosstraining

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CAFMONO supplementation (Active Comparator): The experimental procedure for each participant assume random blind acute ingestion of CAFMONO in individual dose providing 3mg/kg BM of CAF at one of the study visits, which will be separated from other study visits with 7-days wash-out. The preparation will be provided in the form of powder and the individual doses of CAFMONO will be dissolved in 200 mL of water. The test preparation will be ingested within up to 5 minutes. The ingestion will take place 60 minutes before the test exercise.
  Interventions: Dietary Supplement: CAFMONO supplementation
- CAFMIPS_1 supplementation (Active Comparator): The experimental procedure for each participant assume random blind acute ingestion of CAFMIPS_1 in individual dose providing 3mg/kg BM of CAF at one of the study visits, which will be separated from other study visits with 7-days wash-out. The preparation will be provided in the form of powder and the individual doses of CAFMIPS_1 will be dissolved in 200 mL of water. The test preparation will be ingested within up to 5 minutes. The ingestion will take place 60 minutes before the test exercise.
  Interventions: Dietary Supplement: CAFMIPS_1 supplementation
- CAFMIPS_2 supplementation (Active Comparator): The experimental procedure for each participant assume random blind acute ingestion of CAFMIPS_2 in individual dose providing 3mg/kg BM of CAF at one of the study visits, which will be separated from other study visits with 7-days wash-out. The preparation will be provided in the form of powder and the individual doses of CAFMIPS_2 will be dissolved in 200 mL of water. The test preparation will be ingested within up to 5 minutes. The ingestion will take place 60 minutes before the test exercise.
  Interventions: Dietary Supplement: CAFMIPS_2 supplementation
- Placebo treatment (Placebo Comparator): The experimental procedure for each participant assume random blind acute ingestion of placebo (PLA) at one of the study visits, which will be separated from other study visits with 7-days wash-out. The PLA preparation will be provided in the form of powder and dissolved in 200 mL of water. PLA will be ingested within up to 5 minutes. The ingestion will take place 60 minutes before the test exercise.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: CAFMONO supplementation — CAFMONO supplementation - random blind acute intake of in individual dose providing 3mg/kg BM of CAF.
  CAFMONO - Caffeine (anhydrous caffeine), Ostrovit Sp. z o.o., Zambrów, POLAND
  Arms: CAFMONO supplementation
Dietary Supplement: CAFMIPS_1 supplementation — CAFMIPS_1 supplementation - random blind acute intake of in individual dose providing 3mg/kg BM of CAF.
  CAFMIPS_1 - Olimp Redweiler, Olimp Laboratories Sp. z o.o., Dębica, POLAND
  CAFMIPS_1 - Olimp Redweiler, Olimp Laboratories Sp. z o.o., Dębica, POLAND
  Arms: CAFMIPS_1 supplementation
Dietary Supplement: CAFMIPS_2 supplementation — CAFMIPS_2 supplementation - random blind acute intake of in individual dose providing 3mg/kg BM of CAF.
  CAFMIPS_2 - Muscle Clinic Furious, Noblepharma UG, BerlinVertrieb, GERMANY.
  Arms: CAFMIPS_2 supplementation
Dietary Supplement: Placebo treatment — Placebo treatment - random blind acute intake of placebo preparation. Placebo will match the remaining test preparations with taste, colour and consistency, however it will be free of caffeine and any other substances possessing ergogenic potential.
  Arms: Placebo treatment

SUMMARY:
The study aims at assessing the relation between caffeine (CAF) and paraxanthine (PAX) kinetics after acute ingestion of caffeine (3 mg/kg body mass) in the form or mono- or multi-ingredient preparations and CrossFit®-specific performance or selected indicators of psychophysiological state. Blood indicators of muscle damage/recovery, acid-base balance and electrolytes levels will be evaluated. The impact of genetic variations in the polymorphisms rs5751876 in ADORA2A gene and rs762551 in CYP1A2 on CAF/PAX kinetics will be considered.

DETAILED DESCRIPTION:
The main aim of the project is to assess blood and saliva kinetics of CAF and PAX after acute ingestion of caffeine (3 mg/kg body mass) in the form of mono-ingredient preparation (CAFMONO) or two different multi-ingredient pre-workout supplements (CAFMIPS_1 CAFMIPS_2) compared to Placebo (PLA). The impact of CAF/PAX kinetics on CrossFit®-specific performance (as measured via the Fight Gone Bad test <FGB>) and selected psychophysiological indicators such as reaction time, postural stability, the level of focus, alertness, fatigue and feeling of 'energy', as well as the rate of perceived exertion (RPE) will be evaluated. Additionally, blood indicators of muscle damage/regeneration (haematological evaluation; activity of: creatine kinase <CK>, lactate dehydrogenase <LDH>, aspartate aminotransferase <AspAT> and alanine aminotransferase <AlAT>; levels of creatinine <Cre> and mioglobin), acid-base balance (pH, levels of: bicarbonate, , lactate <La>, anion gap; base excess, H+) and concentrations of electrolytes (Ca2+, Na+, K+, Cl-) will be evaluated. Saliva and blood parameters will be assessed before the test preparations ingestion (-10minINT), after ingestion (+15, +30, +45, +60 minINT) and after FGB (+3, +10 minFGB). The indicators of psychophysiological state will be evaluated at -10minINT, +30, +60 minINT, +10minFGB.

The study is a double-blind, randomized, placebo-controlled, cross-over trial. The study consists of preliminary meeting with research team (familiarization with study protocol) and five study visits (T0 - T4), of which T0 is a BLANK visit with no supplementation and supplementation visits (T1 - T4). The testing days will be separated with 7-days wash-out. Investigators aimed to recruit 25 male CrossFit®-trained participants. Random allocation of participants to supplementation order (PLA, CAFMONO, CAFMIPS_1 CAFMIPS_2) will be done using a random sequence generator, with participants being equalised by fat-free mass and number of repetitions in FGB test (established at BLANK visit).

At the preliminary (familiarization) visit the written informed consent for participation in the study protocol will obtained from all participants. After that, anthropometric measurements and familiarization with exercise test procedures (Fight Gone Bad test) will be performed. The biological samples for evaluation of polymorphisms rs5751876 in ADORA2A gene and rs762551 in CYP1A2 will be obtained. At the BLANK visit (T0) no supplementation will be provided. However, the remaining study procedures (anthropometric measurements, blood and saliva collection, FGB and psychophysiological evaluation) will be performed. After the completion of T0 visit, the participants will be randomly assigned to the order of supplementation.

Each of T1-T4 visits will start with body mass and body composition evaluation (electric bioimpedance method). Then the baseline (resting) blood and saliva samples, as well as psychophysiological evaluation will be done (-10minINT). Ten minutes after the baseline evaluation, each participant will ingest the individualized dose of PLA or CAFMONO or CAFMIPS_1/CAFMIPS_2. The doses of the test preparations will be adjusted so that they will provide 3 mg/kg BM of CAF (apart from PLA, which will be taste- and colour-matched but caffeine-free preparation). Sixty-minutes after test preparations ingestion, participants will perform the test exercise - FGB. FGB test comprised of three rounds of five exercises: wall ball, sumo deadlift high pulls, box jump, push press and rowing. Participants are obligated to complete as many repetitions as possible in one minute at each station prior to moving to the next station. After completing each of the five stations, participants will have one minute of rest. The total time to complete FGB test will be17 minutes. After the test preparations intake, before and after FGB the blood and saliva samples drawn, and evaluation of indicators of psychophysiological state will be performed according to the schedule mentioned above.

After collection all the data, comparisons between supplementation treatment conditions (BLANK, PLA, CAFMONO, CAFMIPS_1, CAFMIPS_2) will be performed using repeated measurements analysis of variance (RM ANOVA). Additional models considering gene polymorphisms or treatment order will also be analysed. The level of significance adopted will be p <0.05. Statistical analysis will be performed using Statistica v. 13.3, StatSoft Polska Sp. z o.o., 2022. G*Power software (version 3.1.9.4, Universitat Dusseldorf, Germany) was used to calculate sample size required to obtain a power of approximately 80% (α = 0.05) and large effect size partial eta squared 0.14 in RM ANOVA within factors. Analysis indicated that a sample size of 9 is suitable for detecting differences between five measurements. To account for possible drop-out, the sample size at 25 is established.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from all participants before the study,
* a current medical clearance to practice sports,
* training experience any sport discipline ≥ 5 years and training experience in HIFT ≥ 2 years,
* performing ≥3 training units per week,
* participating in CrossFit® competitions at least once a year.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol,
* serious disease or metabolic problems,
* smoking and tobacco use,
* presence of infectious disease in the previous 4 weeks of the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-07-29 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on discipline-specific performance | 60 minutes after ingestion of tested supplements/placebo
  Total number of repetitions in Fight Gone Bad test and number or repetitions in rounds 1 - 3

SECONDARY OUTCOMES:
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on blood and saliva caffeine and its metabolites levels | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  Blood and saliva CAF and PAX concentrations (µmol/L)
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on reaction time | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  Reaction time (s)
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on postural stability | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  CoP sway area (mm2)
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on subjective levels/feelings of "energy", alertness, focus, fatigue | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  Likert scale 1 - 5
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on the Rate of Perceived Exertion (RPE) | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  RPE evaluated via Borg scale (units: 6 - 20)
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on selected blood markers | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  Blood bicarbonate (mmol/L), lactate (mmol/L), anion gap (mmol/L), H+ (mmol/L), base excess (mmol/L), creatinine (mmol/L), and myoglobin (mmol/L), electrolytes [Ca2+, Na+, K+, Cl-] (mmol/L)
The effect of acute ingestion of the same dose of caffeine (3 mg/kg BM) in form of 3 different preparations on blood indicators of muscle damage/recovery | Pre-ingestion and within 90 minutes after ingestion of tested supplements/placebo
  Activity of creatine kinase (U/L), lactate dehydrogenase (U/L), aspartate aminotransferase (U/L), alanine aminotransferase (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, Prof., PhD, Study Chair — Department of Sports Dietetics, Poznan University of Physical Education; Paulina M Nowaczyk, PhD, Principal Investigator — Department of Sports Dietetics, Poznan University of Physical Education
Locations (1):
- Department of Sports Dietetics, Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided